CLINICAL TRIAL: NCT05326035
Title: A Phase I/II Clinical Study of WJ05129 Tablets in Patients With Locally Advanced or Metastatic Malignant Solid Tumors
Brief Title: A Study of WJ05129 in Advanced Malignant Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The sponsor terminated the study on the basis of the current data and the company's research and development strategy
Sponsor: Suzhou Junjing BioSciences Co., Ltd. (Industry)
Collaborators: Sponsor GmbH (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JS112-001-I
Record Dates: First submitted 2022-02-23; First posted 2022-04-13 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Locally Advanced or Metastatic Malignant Solid Tumors
MeSH Terms: interventions — Paclitaxel

STUDY DESIGN:
Masking Description: None (Open Label)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WJ05129 tablets (Experimental)
  Interventions: Drug: WJ05129
- WJ05129 combined with paclitaxel (Experimental)
  Interventions: Drug: WJ05129; Drug: Paclitaxel injection

INTERVENTIONS:
Drug: WJ05129 — Twice daily (except for single dose), 12 hours apart, fixed time is recommended
Drug: Paclitaxel injection — 80mg/m2 (The maximum dose is 80mg/m2 , and the dose can be adjusted according to the actual situation), The medication is administered on days 1, 8, and 15, and a 28-day period constitutes one cycle.
  Arms: WJ05129 combined with paclitaxel

SUMMARY:
This study was an open, multicenter Phase I/II clinical study of WJ05129 in patients with locally advanced or metastatic malignant solid tumors in China, which was divided into three stages: Single-dose escalation,Combined dose extension and efficacy extension. The study included screening, treatment and follow-up periods. The starting dose of this dose-escalation study was set at 2.5 mg/day. Five dose levels were preset.A more flexible "BOIN" dose escalation method was adopted. The maximum tolerated dose observation period was the first treatment cycle of single administration and multiple consecutive administrations (a total of 2 days) + 21 days = 23 days; In this stage, the two dosage levels of the injectable WJ05129 (RP2D dosage and the lower dose before RP2D) will be selected as the escalating doses for the combined use of WJ05129. The "BOIN" design will be adopted for dose escalation. Paclitaxel 80mg/m2 will be intravenously infused on days 1, 8, and 15. A 28-day cycle will be used, with the first cycle being the DLT observation period.Efficacy expansion phase: It is preliminarily planned to expand three cohorts of Rb negative TNBC and SCLC andOther solid tumors（Such as gastric and esophageal adenomas, gynecological tumors, etc.）, and recruit about 20-40 people in each cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to participate in the clinical trial of this drug, able to understand and sign informed consent, willing and able to comply with the planned visit and study procedures;
2. Age ≥18 to 75 years old, male and female;
3. Locally advanced (except for patients who can be treated with radical therapy) or metastatic malignant solid tumors confirmed by histology or cytology;
4. The single-dose escalation phase requires patients who have failed standard treatment, are intolerant to standard treatment, or have no standard treatment options；The combined dose escalation phase and the efficacy expansion phase require no treatment with taxane drugs for metastatic diseases, with no more than 4 lines of treatment, and meet one of the following conditions:

   1. SCLC: After receiving a platinum-based standard chemotherapy regimen for first-line treatment, whether in localized stage (LS) or extensive stage (ES), there has been progression;
   2. TNBC: After receiving first-line standard treatment, previous adjuvant taxane treatment is allowed, provided that the disease-free interval from (new) adjuvant chemotherapy to the development of metastatic disease is ≥ 1 year;
   3. Other solid tumors: After receiving the first-line standard treatment recommended by CSCO or NCCN guidelines;
5. Eastern Cooperative Oncology Group (ECOG) Physical status score (Annex 2) 0 to 1;
6. Expected survival ≥ 12 weeks;
7. According to the Response evaluation criteria in solid Tumors (RECIST) 1.1 (Annex 4), there is at least one measurable lesion（Applicable only to the dose escalation and efficacy expansion phases of the combination treatment.）;
8. Voluntarily and informed consent to provide fresh biopsy samples before treatment. For patients unable to provide fresh biopsy samples before treatment, archived samples within 2 years can be provided (dose escalation stage is optional, dose expansion and efficacy expansion stage is mandatory);
9. Have sufficient important organ functions, and meet the following standards in laboratory examination ≤ 7 days before the first drug administration:

   A: Blood system (transfusion and cytokine support therapy are not allowed within 14 days prior to initial administration) :
   * Hemoglobin ≥ 90 g/L;
   * Platelet count ≥ 100×109/L;
   * Absolute neutrophil count ≥ 1.5×109/L

   B: Kidney function:
   * Serum albumin ≥30g/L. (Albumin infusion is not allowed within 14 days before administration)
   * Aspartate aminotransferase (AST)/Alanine aminotransferase (ALT) ≤ 2.5 × Upper limit of normal (ULN); If liver metastasis occurred, AST/ALT ≤ 5 × ULN;
   * Serum total bilirubin ≤ 1.5 × ULN; TBIL≤3×ULN in patients with liver metastasis or Gilbert syndrome;
   * Serum creatinine (Cr) ≤1.5 TIMES ULN or creatinine clearance (calculated using the Cockcroft and Gault formula [Appendix 1]) ≥ 50 mL/min;

   C: Coagulation function:

   International standardized ratio (INR), prothrombin time (PT) and activated partial thrombin time (aPTT) ≤ 1.5ULN for patients who did not receive anticoagulant therapy; For those receiving anticoagulant therapy (e.g., low molecular weight heparin or warfarin), the anticoagulant dose should be stable for at least 4 weeks without dose adjustment;

   D: Cardiovascular System:

   According to Fridericia's standard, the QTc interval for males is ≤ 450 ms, and for females it is ≤ 470 ms;
10. A pregnancy test must be performed within 7 days before the first use of the study drug for premenopausal women who are likely to have children. The blood pregnancy test must be negative and must be non-lactation; All enrolled patients (male or female) should take adequate contraceptive measures throughout the treatment period and within 3 months after the end of treatment;

Exclusion Criteria:

1. Persons already known to be allergic to the active ingredients or excipients of the study drugs (WJ05129 tablets) ；
2. Patients previously treated with AURORA A kinase inhibitors (Alisertib, LY3295668, etc.) ；
3. Subjects who received a potent cytochrome CYP3A inhibitor or inducer within 14 days prior to initial administration and who needed to take these drugs throughout the study period;
4. Participate in other clinical studies within 4 weeks prior to initial administration, except during the follow-up period of observational (non-interventional) clinical studies or interventional studies;
5. Inability to swallow drugs orally, or having a condition that seriously affects gastrointestinal absorption as judged by the investigator;
6. Pregnant or lactating women;
7. Two or more malignancies within 5 years prior to first administration. Except for early stage malignant neoplasms (carcinoma in situ or stage I neoplasms) that have been eradicated, such as adequately treated carcinoma in situ of the cervix, basal cell or squamous cell carcinoma, etc.;
8. Underwent major surgery (as determined by the investigator) or was undergoing surgical recovery within 4 weeks prior to initial dosing. Anti-tumor chemotherapy (eluting for 6 weeks for the last chemotherapy with nitrosourea or mitomycin), radiotherapy, targeted therapy, hormone therapy, immunotherapy, or biotherapy within 4 weeks prior to initial administration. Receive anti-tumor or immunomodulatory TCM or Chinese adult medicine preparations within 2 weeks before the first administration;
9. Patients with symptoms of central nervous system metastasis (if asymptomatic and not currently receiving corticosteroid treatment, they are allowed to be enrolled) or primary tumor disease of the central nervous system;
10. Spinal cord compression that cannot be treated radically by surgery and/or radiotherapy, or for previously diagnosed spinal cord compression that is treated without clinical evidence of disease stability ≥1 week prior to randomization;
11. No remission of toxicity after previous antitumor therapy, i.e., no regression to the level specified in baseline, nCI-CTCAE5.0 level 0~1 (except hair loss), or inclusion/exclusion criteria. Irreversible toxicity not reasonably expected to be aggravated by the study drug (e.g., hearing loss) may be included after consultation with the medical monitor ;
12. Repeated drainage is required for third space effusion with clinical symptoms, such as pericardial effusion, pleural effusion and abdominal effusion that cannot be controlled by drainage or other treatment;
13. Patients with active hepatitis B (chronic or acute, defined as patients with HBsAg positive at baseline and HBV DNA copy number greater than the upper limit of the normal value in the laboratory of the study center), or HCV positive (HCV Ab positive and HCV RNA positive);

    1. Patients with prior HBV infection or cured hepatitis B (defined as HBcAb positive and HBsAg negative) can be enrolled. These patients should be tested for HBV DNA expression at the same time before randomization, and the copy number of HBV DNA should be lower than the upper limit of the normal value in the laboratory department of the research center.
    2. Patients with POSITIVE HCV antibodies can only be enrolled if HCV RNA PCR test results are negative.
14. Known human immunodeficiency virus (HIV) positive persons;
15. Active tuberculosis patients;
16. Suffering from other serious complications (such as uncontrollable infection, uncontrollable hypokalemia, hypomagnesia, hypocalcemia, hypertension and thromboembolic diseases, etc.);
17. The patient has a history of major upper gastrointestinal surgery, active gastrointestinal disease or other diseases that may significantly affect drug absorption, metabolism or excretion;
18. Patients with grade 2 or more neuropathy;
19. Have a history of serious cardiovascular disease, including but not limited to: myocardial infarction or cerebrovascular accident within 6 months before enrollment, New York Cardiology > class II congestive heart failure, unstable angina pectoris, arrhythmia, etc.;
20. Prior allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
21. Receive live or attenuated live vaccine within 30 days of initial administration, or plan to receive live vaccine during the study period;
22. Mental illness, alcohol, drug or substance abuse are known;
23. As determined by the investigator, the subject has other factors that may lead to the termination of the study, such as non-compliance with the protocol, other serious diseases requiring combined treatment, serious abnormal laboratory examination, family or social factors, etc., which may affect the safety of the subject, or the collection of data and samples;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2023-12-26 (Actual); Study Completion 2023-12-26 (Actual)

PRIMARY OUTCOMES:
DLT | 2 years
  It is suitable for dose escalation .DLT is defined as any of AE that SMC considers to have occurred during the DLT observation period and may be causally related to WJ05129 and meet DLTcriteria.
The incidence of adverse events (AE) and serious adverse events (SAE) were assessed | 2 years
  It is suitable for dose escalation and dose extension.Incidence and severity of adverse events (AE) and serious adverse events (SAE) as assessed according to NCI-CTCAE 5.0, as well as abnormalities in physical examination, ECOG score, vital signs, electrocardiogram, ophthalmic tests and laboratory tests.
MTD | 2 years
  Defined as the dose level at which the estimated toxicity probability is closest to the target toxicity probability during the DLT observation period
RP2D | 2 years
  RP2D will be determined based on a combination of safety, tolerability, PK and/or pharmacodynamic studies .
Incidence of Treatment-Emergent Adverse Events | 2 years
  Incidence and severity of adverse events (AE) and serious adverse events (SAE) as assessed according to NCI-CTCAE 5.0, as well as abnormalities in physical examination, ECOG score, vital signs, electrocardiogram, ophthalmic tests and laboratory tests.
ORR | 2 years
  It is suitable for the curative effect development stage.Objective Response Rate by RECIST 1.1.

SECONDARY OUTCOMES:
Cmax | 2 years
  Maximum Plasma Concentration
Tmax | 2 years
  It is suitable for dose escalation and dose extension.Time to Cmax
AUC0-t | 2 years
  It is suitable for dose escalation and dose extension.Area under the concentration versus time curve from time 0 to the last measurable concentration
AUC0-inf | 2 years
  It is suitable for dose escalation and dose extension.AUC from time 0 to infinity
t1/2 | 2 years
  It is suitable for dose escalation and dose extension.Elimination half life time
CL/F | 2 years
  It is suitable for dose escalation and dose extension.Clearance
Vd/F | 2 years
  It is suitable for dose escalation and dose extension.Apparent volume of distribution
λz | 2 years
  It is suitable for dose escalation and dose extension.elimination rate constant
DOR | 2 years
  Duration of response
DCR | 2 years
  Disease Control Rate
PFS | 2 years
  Progression-free survival
OS | 2 years
  Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Institute & Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No